CLINICAL TRIAL: NCT00015925
Title: Phase I Clinical-Labratory Study of the Histone Deacetylase (HDA) Inhibitor MS-275 in Adults With Refractory and Relapsed Hematologic Malignancies
Brief Title: MS-275 in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068574, J0253; U01CA069854 (NIH); P30CA006973 (NIH); JHOC-J0253; MSGCC-0050; NCI-2791
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Leukemia; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: refractory multiple myeloma; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; adult acute promyelocytic leukemia (M3); refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Leukemia; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Promyelocytic, Acute; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Congenital Abnormalities | interventions — entinostat

INTERVENTIONS:
Drug: entinostat

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of MS-275 in treating patients who have hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxic effects and pharmacokinetics of MS-275 in patients with poor-risk hematologic malignancy.
* Determine whether this drug induces changes in hematologic differentiation, in terms of changes in morphology, cell surface marker expression, and acetylation status, in these patients.
* Determine whether this drug induces clinical response in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive oral MS-275 on days 1, 8, 15, and 22. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of MS-275 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 25-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following histologically confirmed diagnoses:

  * Acute myeloid leukemia (AML)

    * Newly diagnosed de novo AML in patients over 60 years old with the following poor-risk features:

      * Antecedent hematologic disorder
      * Complex karyotype or other adverse cytogenetics
      * Stem cell immunophenotype
    * AML arising from myelodysplastic syndromes (MDS)
    * Secondary AML
    * Relapsed or refractory AML, including primary induction failure
  * MDS

    * Poor-risk, defined as the following:

      * International Performance Score at least 1.5
      * More than 10% marrow blasts
      * Cytopenias in at least 2 lineages
    * Refractory anemia with excess blasts (RAEB)
    * RAEB in transformation
    * Chronic myelomonocytic leukemia
  * Acute lymphoblastic leukemia (ALL)

    * Newly diagnosed de novo ALL in patients over 60 years old with the following poor-risk features:

      * Complex karyotype or other adverse cytogenetics
      * Mixed lineage immunophenotype
    * Relapsed or refractory ALL, including primary induction failure
  * Chronic myelogenous leukemia (CML)

    * CML in accelerated phase or blast crisis
    * Interferon-refractory CML in chronic phase
  * Multiple myeloma (MM)

    * Relapsed or refractory, including prior autologous stem cell transplantation
  * Acute promyelocytic leukemia

    * Prior treatment with tretinoin
    * Ineligible for arsenic trioxide
    * No evidence of active coagulopathy
    * Low-risk for developing clinically significant coagulopathy during study

      * Low tumor burden by marrow aspiration at time of relapse
      * No prior coagulation-related sequelae (deep vein thrombosis, pulmonary embolism, or CNS thrombosis or bleed)
* Failure after primary induction therapy or relapse after complete remission allowed if patient received no more than 3 courses of prior induction/reinduction therapy
* Not eligible for curative stem cell transplantation
* No hyperleukocytosis with at least 50,000/mm^3 leukemic blasts
* No active CNS leukemia
* No plasma cell leukemia
* No amyloidosis resulting in major organ dysfunction

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics
* No disseminated intravascular coagulation
* No hyperviscosity

Hepatic:

* AST/ALT no greater than 2 times normal
* Alkaline phosphatase no greater than 2 times normal
* Bilirubin no greater than 1.5 times normal

Renal:

* Creatinine no greater than 1.5 times normal
* No uncorrected hypercalcemia

Cardiovascular:

* See Disease Characteristics
* LVEF at least 45% by MUGA or echocardiogram
* No intrinsic impaired cardiac function, including any of the following:

  * Myocardial infarction within the past 3 months
  * Prior severe coronary artery disease
  * Cardiomyopathy
  * Congestive heart failure

Other:

* No active uncontrolled infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 1 week since prior growth factors (epoetin alfa, filgrastim [G-CSF], sargramostim [GM-CSF], interleukin [IL]-3, or IL-11)
* At least 4 weeks since prior autologous stem cell transplantation
* No prior allogeneic stem cell transplantation
* No concurrent immunotherapy

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy and recovered
* At least 24 hours since prior hydroxyurea or mercaptopurine for prevention of leukostasis
* No concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 2 weeks since prior emergency radiotherapy to large soft tissue or lytic bony lesions for MM
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* At least 24 hours since other prior noncytotoxic agents for prevention of leukostasis
* No other concurrent antitumor therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-02

CONTACTS AND LOCATIONS:
Overall Officials: Judith E. Karp, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland